CLINICAL TRIAL: NCT05608720
Title: Randomized Clinical Trial to Test a Preparation Protocol for the First Pediatric Dental Visit.
Brief Title: Preparation Protocol for the First Pediatric Dental Visit
Acronym: PREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Simone Bagattoni, Principal investigator, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: bagattoni1
Record Dates: First submitted 2022-10-27; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Behavior, Child; Dentist-Patient Relations
Keywords: behavior management; first dental visit
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Information Booklet prior to the dental visit
  Interventions: Behavioral: Information Booklet
- control group (No Intervention): no information prior to the dental visit

INTERVENTIONS:
Behavioral: Information Booklet — Information Booklet prior to the dental visit
  Arms: study group

SUMMARY:
To date, not enough attention has been paid to the role of communication before the first dental visit to encourage the child's cooperation and avoid dysfunctional behaviors. The dentist can provide parents with the information they need to adequately prepare the child for treatment. The present study aims to investigate the effectiveness of an infor-mation booklet to promote pediatric patients' cooperation during the first dental visit

DETAILED DESCRIPTION:
The aim of the study was to test an Information Booklet preparing the child to the first dental vis-it. Forty-five children and one parent per included child took part in the trial. Children were ran-domized in two groups: the Information Booklet was e-mailed to the parents of the study group. At the end of the visit, the dentist and the parent evaluated the child's behavior through the Frankl Behavior Rating Scale (FBRS) and the utility of the Booklet through a Likert scale. The children evaluated the pleasantness of the visit and the perceived pain through the Wong-Baker FACES® Pain Rating Scale (WBFPRS).

ELIGIBILITY:
Inclusion Criteria:

* child requiring a first dental visit

Exclusion Criteria:

* previous dental visits, intellectual disability, mother tongue other than Italian, una-vailable e-mail address

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
child's behavior assessed by dentist with the Frankl Behavior Rating Scale (FBRS) | immediately after the intervention
  FBRS: values from 1 (Definitely negative) to 4 (definitely positive)

SECONDARY OUTCOMES:
self reported pain assessed by the Wong Baker faces pain rating scale (WBFPRS) | immediately after the intervention
  WBFPRS: from 0 (no hurt) to 10 (hurts worst)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Bagattoni, Principal Investigator — Bologna University
Locations (1):
- Servizio di Assistenza Odontoiatrica per disabili in età evolutiva e di odontoiatria infantile, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No